CLINICAL TRIAL: NCT04825873
Title: The Observational Safety Study for Nivolumab in China Routine Oncology Practice
Brief Title: A Study to Assess Safety of Nivolumab in Routine Oncology Practice in China
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-8JH
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Non-Small Cell Lung Cancer; Squamous Cell Carcinoma of Head and Neck
Keywords: BMS-936558; China; Nivolumab; Non-Small Cell Lung Cancer; Platinum-based chemotherapy; Postmarketing observational study; Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (4):
- Cohort 1: Prospective observation of participants with non-small cell lung cancer (NSCLC)
- Cohort 2: Prospective observation of participants with squamous cell carcinoma of head and neck (SCCHN)
- Cohort 3: Retrospective observation of participants with NSCLC
- Cohort 4: Retrospective observation of participants with SCCHN

SUMMARY:
The purpose of this study is to assess the safety of nivolumab in routine cancer practice in China. Part one of the study will investigate nivolumab for non-small cell lung cancer previously treated with platinum-based chemotherapy that has locally advanced or has spread. Part two will investigate nivolumab for post-platinum squamous cell carcinoma of head and neck that is recurrent or has spread. Part three will investigate nivolumab for locally advanced or metastatic non-small cell lung cancer. Part four will investigate nivolumab for recurrent or metastatic squamous cell carcinoma of head and neck.

ELIGIBILITY:
Inclusion Criteria:

Part 1

* Histologically or cytologically confirmed diagnosis of locally advanced/metastatic non-small cell lung cancer (NSCLC) participants
* Treatment with nivolumab per physician's prescription

Part 2

* Histologically or cytologically confirmed diagnosis of recurrent/metastatic squamous cell carcinoma of head and neck (SCCHN)
* Treatment with nivolumab for recurrent or metastatic SCCHN

Part 3

* Histologically or cytologically confirmed diagnosis of locally advanced/metastatic NSCLC
* Participants with at least one dose of nivolumab administered since June 2018

Part 4

* Histologically or cytologically confirmed diagnosis of recurrent/metastatic SCCHN
* Participants with at least one dose of nivolumab administered since September 2019

Exclusion Criteria:

* Prior participation in a clinical trial within the past 4 weeks
* Current or pending participation in a clinical trial
* Current or pending systemic treatment for cancer other than NSCLC for part 1 and SCCHN for part 2
* Previously treated with immune checkpoint inhibitors for part 3 and part 4
* Participants must not have any other concurrent primary tumor(s) for part 3 and part 4

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In part 1 and part 3, the study population consists of adults with locally advanced or metastatic NSCLC treated with nivolumab per physician's prescription.
  In part 2 and 4, the study population consists of adults with recurrent or metastatic SCCHN who are treated with nivolumab per physician's prescription.
Sampling Method: Non-Probability Sample
Enrollment: 3102 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Incidence rate of nivolumab-related immune-related adverse events (irAEs) | Up to approximately 48 months
Severity of nivolumab-related irAEs | Up to approximately 48 months
Incidence rate of nivolumab-related adverse events (AEs) | Up to approximately 48 months
Severity of nivolumab-related AEs | Up to approximately 48 months
Incidence rate of nivolumab-related serious adverse events (SAEs) | Up to approximately 48 months
Severity of nivolumab-related SAEs | Up to approximately 48 months
Incidence rate of treatment-related adverse events TRAEs | Up to approximately 48 months
  Part 3 and Part 4
Severity of TRAEs | Up to approximately 48 months
  Part 3 and Part 4
Management of irAEs | Up to approximately 48 months
  Part 3 and Part 4
Distribution of outcomes of irAEs | Up to approximately 48 months
  Part 3 and Part 4

SECONDARY OUTCOMES:
Management of Common Terminology Criteria for Adverse Event (CTCAE) Grades 2-5 nivolumab-related irAEs | Up to approximately 48 months
Management of CTCAE Grades 2-5 nivolumab-related AEs | Up to approximately 48 months
  Part 1 and Part 2
Management of CTCAE Grades 2-5 nivolumab-related SAEs | Up to approximately 48 months
  Part 1 and Part 2
Distribution of outcomes of CTCAE Grades 2-5 irAEs associated with nivolumab when managed according to the risk management algorithms described in the nivolumab label | Up to approximately 48 months
  Part 1 and Part 2
Distribution of outcomes of CTCAE Grades 2-5 AEs associated with nivolumab when managed according to the risk management algorithms described in the nivolumab label | Up to approximately 48 months
  Part 1 and Part 2
Distribution of outcomes of CTCAE Grades 2-5 SAEs associated with nivolumab when managed according to the risk management algorithms described in the nivolumab label | Up to approximately 48 months
  Part 1 and Part 2
Distribution of treatment patterns of nivolumab in routine oncology practice: Treatment duration | Up to approximately 48 months
  Part 1 and Part 3
Distribution of treatment patterns of nivolumab in routine oncology practice: Treatment sequencing | Up to approximately 48 months
  Part 1 and Part 3
Distribution of treatment patterns of nivolumab in routine oncology practice: Reasons for nivolumab discontinuation | Up to approximately 48 months
  Part 1 and Part 3
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Age | Up to approximately 48 months
  Part 1
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Sex | Up to approximately 48 months
  Part 1
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Weight | Up to approximately 48 months
  Part 1
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Height | Up to approximately 48 months
  Part 1
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: BMI | Up to approximately 48 months
  Part 1
Distribution of clinical characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Smoking status | Up to approximately 48 months
  Part 1
Distribution of clinical characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Eastern Cooperative Oncology Group (ECOG) performance status | Up to approximately 48 months
  Part 1
Distribution of clinical characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Comorbidities | Up to approximately 48 months
  Part 1
Distribution of clinical characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Disease history | Up to approximately 48 months
  Part 1
Distribution of clinical characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Treatment history | Up to approximately 48 months
  Part 1
Distribution of treatment outcomes of NSCLC participants treated with nivolumab from start of nivolumab treatment: overall survival (OS) | Up to approximately 48 months
  Part 1 and Part 3
Distribution of treatment outcomes of NSCLC participants treated with nivolumab from start of nivolumab treatment: real-world progression free survival (rwPFS) | Up to approximately 48 months
  Part 1 and Part 3
Distribution of treatment patterns of nivolumab for recurrent squamous cell carcinoma of head and neck (SCCHN) | Up to approximately 48 months
  Part 2 and Part 4
Distribution of treatment patterns of nivolumab for metastatic SCCHN | Up to approximately 48 months
  Part 2
Distribution of demographic characteristics of SCCHN participants treated with nivolumab at initiation of nivolumab treatment: Age | Up to approximately 48 months
  Part 2
Distribution of demographic characteristics of SCCHN participants treated with nivolumab at initiation of nivolumab treatment: Sex | Up to approximately 48 months
  Part 2
Distribution of demographic characteristics of SCCHN participants treated with nivolumab at initiation of nivolumab treatment: Weight | Up to approximately 48 months
  Part 2
Distribution of demographic characteristics of SCCHN participants treated with nivolumab at initiation of nivolumab treatment: Height | Up to approximately 48 months
  Part 2
Distribution of demographic characteristics of SCCHN participants treated with nivolumab at initiation of nivolumab treatment: BMI | Up to approximately 48 months
  Part 2
Distribution of demographic characteristics of SCCHN participants treated with nivolumab at initiation of nivolumab treatment: Alcohol consumption | Up to approximately 48 months
  Part 2
Distribution of demographic characteristics of SCCHN participants treated with nivolumab at initiation of nivolumab treatment: Human papillomavirus (HPV) status | Up to approximately 48 months
  Part 2
Distribution of clinical characteristics of SCCHN participants treated with nivolumab at initiation of nivolumab treatment: Smoking status | Up to approximately 48 months
  Part 2
Distribution of clinical characteristics of SCCHN participants treated with nivolumab at initiation of nivolumab treatment: Eastern Cooperative Oncology Group (ECOG) performance status | Up to approximately 48 months
  Part 2
Distribution of clinical characteristics of SCCHN participants treated with nivolumab at initiation of nivolumab treatment: Comorbidities | Up to approximately 48 months
  Part 2
Distribution of clinical characteristics of SCCHN participants treated with nivolumab at initiation of nivolumab treatment: Disease history | Up to approximately 48 months
  Part 2
Distribution of clinical characteristics of SCCHN participants treated with nivolumab at initiation of nivolumab treatment: Treatment history | Up to approximately 48 months
  Part 2
Distribution of treatment effectiveness of SCCHN participants treated with nivolumab from the start of nivolumab treatment: OS | Up to approximately 48 months
  Part 2 and Part 4
Distribution of treatment effectiveness of SCCHN participants treated with nivolumab from the start of nivolumab treatment: rwPFS | Up to approximately 48 months
  Part 2 and Part 4

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- China (2):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Shanghai, Shanghai Municipality

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html